CLINICAL TRIAL: NCT05128084
Title: Platelet Transfusion in Pediatric Heart Surgery and Impact of Amotosalen Treatment
Brief Title: Amotosalen and Platelet Transfusion in Pediatric Heart Surgery
Acronym: TransPédia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7977
Record Dates: First submitted 2021-10-12; First posted 2021-11-19 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-10

CONDITIONS: Congenital Heart Disease in Children
Keywords: Congenital Heart; Platelet transfusion; Procoagulant drugs; Amotosalen; Pediatric heart surgery

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
High level of security during blood transfusion has been achieved by donor selection and pathogen detection using serology or direct identification. Nevertheless, blood banking becomes hazardous during epidemic outbreaks or facing new pathogens. Amotosalen, a psoralen, targets nucleic acids and destroys them after ultraviolet exposure, resulting in inactivation of pathogens.

Treatment inoccuity and efficacy have been demonstrated but preservation of platelet functions after treatment is still debated. Previous studies focused on hematological patients. There is no evidence for an increased requirement of transfused platelets to achieve platelet count target. Studies in heart surgery are lacking.

The investigators perform a multicenter, retrospective, "before/after", controlled study in minor patients requiring heart surgery with cardiopulmonary bypass. One center (Strasbourg) uses Amotosalen-treated platelet concentrates since 2006 (control arm). This treatment becomes available in Bordeaux in October 2017 (intervention arm). There is two periods of inclusion: one "before" (January 2016 to June 2017) and one "after" (January 2018 to June 2019).

ELIGIBILITY:
Inclusion criteria:

* Minor patient (<18 years old)
* Cardiac surgery act under cardiopulmonary bypass for correction of congenital heart disease
* Platelet transfusion for any reason
* Cardiac surgery performed at Bordeaux or Strasbourg University Hospital over two periods:

  * Period A: January 01, 2016 - June 30, 2017 (before treatment)
  * Period B: January 01, 2018 - June 30, 2019 (after treatment)
* Subject (and / or his parental authority) not having expressed, after information, his opposition to the reuse of his data for the purposes of this research

Exclusion criteria

* Subject (and / or his parental authority) having expressed, after information, his opposition to the reuse of his data for the purposes of this research
* Presence or installation of transient circulatory assistance (outside of the CEC) or definitive
* Heart or cardiopulmonary transplantation

Ages: 1 Year to 17 Years | Sex: All
Age Groups: Child
Study Population: Minor patient having had cardiac surgery act under cardiopulmonary bypass for correction of congenital heart disease
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Retrospective study of the non-inferiority of treatment with Amotosalen of platelet concentrates over transfusion during pediatric cardiac surgery | Files analysed retrospectively from January 01, 2016 to June 30, 2019 will be examined]

CONTACTS AND LOCATIONS:
Overall Officials: Xavier DELABRANCHE, MD, Principal Investigator — Service d'Anesthésie et Réanimation chirurgicale - Hôpitaux Universitaires de Strasbourg
Locations (1):
- Service d'Anesthésie et Réanimation chirurgicale - Hôpitaux Universitaires de Strasbourg, Strasbourg, France